CLINICAL TRIAL: NCT05007158
Title: A Prospective Case-control Validation of Procalcitonin as a Biomarker Diagnosing Pacemaker and Implantable Cardioverter Defibrillator Pocket Infection
Brief Title: Validation of Procalcitonin as a Biomarker Diagnosing CDI
Acronym: (DIRT II)
Status: Completed | Type: Observational
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: Sponsor
Other Study IDs: GER-EP-023
Record Dates: First submitted 2021-07-31; First posted 2021-08-16 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2021-07

CONDITIONS: Cardiac Implantable Electronic Device Infections

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- pocket infection: Patients with isolated pocket infection were diagnosed in the presence of local signs of inflammation (one or more of erythema, pain, warmth, swelling, induration, tenderness, or fluctuation), wound dehiscence, hardware protrusion or pus discharge at the pocket in the absence of systemic findings.
  Interventions: Other: procalcitonin blood test
- CIED systemic infection: Patient s with a CIED systemic infection, diagnosed as the presence of pocket infection accompanied by bacteraemia or echocardiographic finding suggestive of infective endocarditis, but not fulfilling the Duke criteria.
  Interventions: Other: procalcitonin blood test
- Lead-associated infective endocarditis: Patients with infective endocarditis, diagnosed according to modified Duke criteria
  Interventions: Other: procalcitonin blood test
- control group: CIED Patients presenting for elective device exchange or planned lead revision between without local or systemic infections were selected as controls
  Interventions: Other: procalcitonin blood test

INTERVENTIONS:
Other: procalcitonin blood test — blood samples of all participants were analyzed for procalitonin levels, using a commercially available procalitonin testing kit

SUMMARY:
Cardiac device infections (CDI), especially pocket infections, are difficult to be diagnosed. Device pocket infections are not associated with elevated white blood cell count. CRP is only assoziated with a low sensitivity. The diagnosis of a local pocket infection is challenging and relies primarily on the clinical presentation. The prospective DIRT study identified procalcitonin (PCT) among 14 biomarkers as the most promising biomarker to aid the diagnosis of pocket infection.

The study aims to validate the proposed PCT cut-off value of 0.05 ng/ml for the diagnosis of pocket infection

ELIGIBILITY:
Inclusion Criteria:

• device associated infections

Exclusion Criteria:

* malignancy
* cytostatic or immunomodulating therapy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients presenting with cardiac device infection CDI
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-12-01 (Actual); Primary Completion 2021-10-10 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
diagnostic value of PCT | pre-intervention/procedure/surgery. i.e. at the time of CIED explantation. Measurement of PCT as an biomarker revealing the acute infection (like a sepsis marker)
  diagnostic value of PCT in differentiating local pocket infection from infection-free controls and calculated the sensitivity and specificity of the pre-established cut-off value of 0.05 ng/ml

IPD SHARING:
Plan to Share IPD: No